CLINICAL TRIAL: NCT00005069
Title: Phase II Trial of Arsenic Trioxide (NSC #706363) in Patients With Advanced Renal Cell Carcinoma
Brief Title: Arsenic Trioxide in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-107; CDR0000067674 (Registry Identifier: PDQ (Physician Data Query)); NCI-T99-0105
Record Dates: First submitted 2000-04-06; First posted 2004-05-26 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of arsenic trioxide in patients with metastatic renal cell cancer. II. Determine the safety of this regimen in this patient population.

OUTLINE: Patients receive arsenic trioxide IV over 1-4 hours daily for 5 days. Treatment continues every 4 weeks for a maximum of 12 courses in the absence of disease progression or unacceptable toxicity. Patients are followed for at least 1 month.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 6-19 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic renal cell cancer Bidimensionally measurable disease No brain metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 70-100% Life expectancy: Greater than 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal ALT or AST no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN (no greater than 1.95 mg/dL at MSKCC) Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 4 months after study No other prior malignancy unless curatively treated and disease free for the past 5 years and considered low risk for recurrence

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy and recovered No concurrent biologic therapy Chemotherapy: At least 4 weeks since prior cytotoxic chemotherapy and recovered No other concurrent cytotoxic chemotherapy Endocrine therapy: At least 4 weeks since prior hormonal therapy and recovered No concurrent hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy No concurrent radiotherapy Surgery: At least 4 weeks since prior major surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States